CLINICAL TRIAL: NCT06787300
Title: The Effect of Stories to Empower Mothers Programme on Postpartum Depression in Primigravid Pregnant Women
Brief Title: Stories That Empower Mothers and Postpartum Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Ege Miray Topcu, research assistant, Ege University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-8T/27
Record Dates: First submitted 2025-01-11; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Postpartum Depression
Keywords: postpartum depression; pschiatric nursing; promotion of mental health; nursing intervention
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: The research is conducted in a non-randomised experimental follow-up research design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SEM (Experimental): these participants are willing to attemp for programme(Stories that Empower Mothers "SEM")
  Interventions: Behavioral: Stories that Empowered Mother
- control group (No Intervention): these participant is control group.this group is expected to complete only the post-test and follow-up tests. Pregnant women will continue routine pregnancy follow-up.

INTERVENTIONS:
Behavioral: Stories that Empowered Mother — this intervention is made by resercher for this research.
  Other Names: Stories that Empower Mothers Programme
  Arms: SEM

SUMMARY:
Postpartum depression is a condition that occurs after birth and is difficult for mothers. Research shows that experiencing postpartum depression once increases the risk of experiencing it in subsequent pregnancies. At the same time, there are findings in the literature that pregnant women with postpartum depression experience mental difficulties, anxiety or depression during pregnancy. For this reason, this study aims to determine the risk of postpartum depression in pregnant women who are pregnant for the first time during pregnancy and to prevent this risk from occurring in the postpartum period. For this purpose, 'Stories to empower mothers' programme was created. This programme was created by researchers who are specialist psychiatric nurses, psychotherapists and art therapists and finalised with expert opinions. The programme consists of six sessions. The sessions are individual and are conducted online except for the first session. A storybook is formed at the end of the programme with the steps followed during the sessions. While creating this storybook, the themes of self-knowledge, defining the situation, identifying difficulties, identifying sources of help, discovering strengths and creating new coping strategies are addressed by using art therapy techniques. The aim of the study is to examine the effect of the 'Stories Empowering Mothers Programme' on the risk of postpartum depression in pregnant women experiencing their first pregnancy.

The research is conducted in a non-randomised experimental follow-up research design. Pregnant women who meet the inclusion criteria of the study can be included in the experimental or control group according to their wishes. The data collection process in the study proceeds in the order of determining the target group, pre-test (24-32nd gestational week), post-test (after 5 weeks), follow-up one test (postpartum 2nd-4th week) and follow-up two tests (postpartum 10th-12th week). The data are obtained with the Case Report Form and Postpartum Information Form prepared by the researcher and EPDI, BDI and Brief Psychological Resilience Scale forms.

Expert support will be obtained for statistical analyses. Ethics committee permission was obtained before the research was started to be conducted. The research is a doctoral thesis supported by TÜBİTAK.

DETAILED DESCRIPTION:
Within the scope of this research, it is aimed to develop the 'Stories that Empower Mothers' programme, which can evaluate the mental health of women from the pregnancy process, based on the basic skills and philosophy of psychiatric nursing, using the therapeutic power of art, and to evaluate the effect of this programme developed within the scope of this doctoral thesis on the risk of postpartum depression and psychological resilience of pregnant women.

The research is a quantitative, non-randomised experimental follow-up study with intervention and control groups. The research was conducted in a pretest, posttest and two follow-up tests for both intervention and control groups.

The population of the study consisted of primigravid women who applied to Ege University Hospital Gynaecology and Obstetrics outpatient clinic. The number of pregnant women applying to Ege University Gynaecology and Obstetrics outpatient clinic is about 60 per day, but it is not known how many of the applications are first pregnancies. The sample selection method was not used in the study, and all pregnant women who met the criteria for inclusion in the study within the specified time interval were included in the experimental or control group according to their preferences. In order to determine the sample size, the power analysis of the study was calculated with the G*Power 3.1.9.7 programme. For the two groups, it was found appropriate to work with a total of 24 people with 80% power and 0.05 error, taking the effect size at a moderate level (f = 0.25). It was planned to study with a total of 30 patients (15 people in each group).

Dependent Variables In the study, women's descriptive characteristics, postnatal evaluations, Beck Depression Scale, Edinburg Postnatal Depression Scale and Psychological Resilience Scale for Adults score levels constitute the dependent variables.

Independent Variables Stories that empower mothers programme is the independent variable. The research data are obtained with the Case Report Form and Postnatal Information Form prepared by the researcher, and EPBS, BDI and Brief Psychological Resilience Scale. Permission for the scales was obtained from the authors via e-mail.

The Stories That Empower Mothers program is planned as a nursing experimental program using art therapy techniques prepared by the researcher. The aim of the program is to reduce the risk of depression in the postpartum period by increasing the psychological resilience of pregnant women whose postpartum depression risks are determined. While structuring the program, it was created by evaluating the sub-concepts of psychological resilience and art therapy techniques within the scope of the psychiatric nursing philosophy and the care standards of the psychiatric nurse. Among the studies examined, it is seen that different branches of art are used in the emotional state of pregnant women and postpartum depression, and it is recommended to use the therapeutic function of art. The program utilizes visual art activities such as imagery, painting, and story writing techniques. The program flow begins with introductions, introducing the program to the pregnant woman, and explaining the program and session goals. It is completed with the discovery of the pregnant women about themselves, their feelings about becoming a mother, their coping mechanisms, their strengths, and their support mechanisms, and the creation of a storybook product from this discovery journey. The general flow of the sessions progresses with the stages of warming up, implementing the application determined for the session, summarizing the session, and planning the next session. After the program was created, it was presented to expert opinion before implementation.

It is seen that the program sessions implemented within the scope of the literature are organized between 6 and 8 weeks .The Stories That Empower Mothers Program coincides with the beginning of the third trimester of pregnant women and is planned as six sessions. The first of the sessions will be held face-to-face with the women in a clinical environment with a pre-test. The other five sessions will be conducted online. Within the scope of the program, visual art materials such as paper, pencil, glue, paint, scissors are used to support the creativity of the pregnant women. The art products are then provided by the researcher, and an additional list of suggestions is provided to the pregnant women in case they want to enrich the session. At the beginning of each session, light music is used in warm-up activities to support the pregnant women to focus on the here and now. The Stories That Empower Mothers Program is carried out through an online and free video call program (Skype). How to set up and use the program is explained to the pregnant women with a visual. No video or audio recordings are made in the program, and this information is explained to the pregnant women at the beginning of each session. The pregnant women are also asked to create an environment that will not interfere with the interview and where they can ensure their own privacy during the interview. At the same time, at the beginning of the session, the researcher shows the pregnant woman the room she is in, indicating that she ensures her privacy. The researcher keeps a report containing her observations about the continuity of the process and the individuals' conditions during and after the sessions, but these reports are not included in the data of the study. At the end of the sessions, the pregnant women are asked to photograph the art products they have created and send them to the researcher. Pregnant women are informed that these photographs will only be used within the thesis and will not be shared in any other virtual environment.

ELIGIBILITY:
Inclusion Criteria:

* First pregnancy,
* Singleton pregnancy,
* Gestational week between 24-32,
* Regular doctor follow-up,
* Scored ≥ 10 on the EDBS,
* Scored < 17 on the BDI,
* Literate,
* No disability in sensory organs that would prevent communication,
* Owning a smart phone or computer,
* Having internet access,
* Volunteering

Exclusion Criteria:

* Being in the first trimester of pregnancy,

  * Being treated/therapized with any psychiatric diagnosis,
  * Having a risky pregnancy,
  * Being at risk of premature birth and developing it,
  * Having any complications related to pregnancy (gestational diabetes, hypertension, bleeding, etc.),
  * The baby is not healthy,
  * Developing complications during and after birth,
  * The baby needs intensive care after birth,
  * Having a baby lost,
  * Having a premature birth (<37 weeks),
  * The mother has experienced serious daily life difficulties (disaster, loss, etc.),
  * Not attending three or more of the six sessions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The study is conducted with primagravida pregnant women.
Enrollment: 30 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-06-10 (Estimated); Study Completion 2025-11-02 (Estimated)

PRIMARY OUTCOMES:
Case Report Form | 24 - 32. gestational week
  The case report form created by the researcher is a form consisting of questions regarding the contact information, age, marital status, pregnancy information, whether the pregnancy was desired, and whether any treatment was received for the pregnancy of the pregnant women participating in the study. The case report form will be applied to all pregnant women in order to determine the sample group.
Edinburgh postpartum depression scale | pre-test( 24 - 32. gestational week), post-test( (30 to 38 weeks of gestation, 6 weeks after the pretest) , follow-up 1 test, (2 - 4. postnatal week), follow-up 2 test (10 -12. postanal week)
  It was developed by Cox et al. in 1987, and its validity and reliability have been tested in many countries and different languages to date, and its validity and reliability study in our country was conducted by Engindeniz et al. (1996). The scale consists of 10 items. The items are evaluated in a 4-point Likert format and are scored between 0-3. The lowest score that can be obtained from the scale is 0, and the highest score is 30. Each item in the scale is evaluated as 0, 1, 2, 3, and the scoring is reversed (3, 2, 1, 0) in the evaluation of items 3, 5, 6, 7, 8, 9, and 10.
Beck Depression Inventory | pre- test( 24 - 32. gestational week),
  eck Depression Inventory is a four-point Likert-type self-assessment scale developed by Beck et al. (1961) to measure the physical, emotional, cognitive and motivational components of depression. The scale is graded between '0-3' and consists of 21 questions. The minimum and maximum values of the scale are 0-63. Although depression is assessed in four degrees on the scale; 5-9 points indicate normal, 10-16 points indicate mild-moderate, 17-29 points indicate moderate-severe and 30-63 points indicate severe depression (Beck et al., 1961). The inventory will be used to support an inclusion-exclusion criterion in determining the target population of the research.
Brief Resilience Scale | pre-test( 24 - 32. gestational week), post-test(30 to 38 weeks of gestation, 6 weeks after the pretest)
  The scale was developed by Smith et al. (2008) to measure the psychological resilience of individuals. KPSS is a 5-point Likert-type, 6-item, self-reporting measurement tool. Items 2, 4 and 6 are reverse coded. KPSS is a 5-point Likert-type scale. It has an answer key of "Not at all appropriate" (1), "Not appropriate" (2), "Somewhat appropriate" (3), "Appropriate" (4), "Completely appropriate" (5). After the reverse coded items in the scale are translated, high scores indicate high psychological resilience.
Postpartum Information Form | Follow-up 1 test, (2 - 4. postnatal week)
  The postpartum interview form is a form that will be applied to both the experimental and control groups after the women give birth. The form evaluates the women's birth dates, birth methods, and whether they received support during the postpartum period.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all IPD collected
Supporting Information: Study Protocol
Time Frame: december 2025 - december 2028

REFERENCES:
- [Result] Perkins R, Yorke S, Fancourt D. How group singing facilitates recovery from the symptoms of postnatal depression: a comparative qualitative study. BMC Psychol. 2018 Aug 17;6(1):41. doi: 10.1186/s40359-018-0253-0. PMID 30119704
- [Result] Demecs IP, Fenwick J, Gamble J. Women's experiences of attending a creative arts program during their pregnancy. Women Birth. 2011 Sep;24(3):112-21. doi: 10.1016/j.wombi.2010.08.004. Epub 2010 Sep 24. PMID 20869936
- [Result] Crane T, Buultjens M, Fenner P. Art-based interventions during pregnancy to support women's wellbeing: An integrative review. Women Birth. 2021 Jul;34(4):325-334. doi: 10.1016/j.wombi.2020.08.009. Epub 2020 Sep 8. PMID 32912739